CLINICAL TRIAL: NCT04385862
Title: The Use of a Continuous Glucose Monitoring System (Dexcom G6) in Hospitalized Patients for Acute Care
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor problem of delivering material
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CGM-SI
Record Dates: First submitted 2020-05-08; First posted 2020-05-13 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2020-05

CONDITIONS: Continuous Glucose Monitoring
Keywords: Continuous glucose monitoring; Intravenous insulin; Diabetes; Insulin; Glucose measurements
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

SUMMARY:
The state of a coronavirus disease pandemic (COVID-19) was declared by the World Health Organization on March 11, 2020. Hospitalized patients receiving intravenous (IV) insulin therapy have been identified in the hospital setting as a group that places health care workers at high risk of contamination. Indeed, the many capillary blood glucose measurements required to adjust the IV insulin doses involve direct contact with the patient. It is generally recommended to measure blood sugar every 1 to 2 hours with an IV insulin infusion. Ensuring a working method allowing optimal monitoring of patients' blood sugar levels while limiting the risk of contamination of health professionals is therefore to be preferred.

Continuous Glucose Monitoring (CGM) systems are minimally invasive devices that allow you to get a blood glucose measurement every 5 to 15 minutes, and some devices allow you to access your blood sugar profile without having to be in contact with the patients. These devices are approved, validated, and widely used in diabetic ambulatory populations. The principle is based on a measurement of glucose in the interstitial fluid under the skin.

DEXCOM G6 is the only device currently approved in Canada that does not require calibration using a capillary blood glucose level or contact with the patient for remote data transmission. A sensor installed on the skin makes it possible to measure blood sugar from the interstitial fluid. A transmitter installed on the sensor sends the data to a receiver which can be remote from the patient (up to 6 meters). Its use in an acute care setting, however, is not approved in Canada. However, Health Canada issued an emergency order on April 25, 2020 allowing the use of Dexcom G6 in hospitals during the COVID-19 pandemic.

The CGM offers several potential advantages compared to the capillary glycemia currently used to ensure the follow-up of insulin-treated patients thanks to the real-time measurement of the glycemia and their transmission at a distance. In intensive care the SGC has the potential:

* For staff to limit contact with patients infected with COVID-19 (reduction in the use of personal protective equipment and contamination) while ensuring close monitoring of blood glucose levels for the adjustment of insulin therapy.
* For patients to reduce the discomfort related to multiple capillary blood sugar levels and possibly better detection of hypoglycaemia

This study is the first step in a 2-phase research program, the ultimate goal of which is to use a CGM to replace capillary blood glucose in hospitals to adjust intravenous (IV) insulin therapy.

The objective of the first study presented in this protocol is to validate the use of a continuous glucose monitoring system (CGM) for glycemic monitoring in patients hospitalized in intensive care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥ 18 years old) admitted to intensive care at the CHUM
* IV insulin infusion scheduled for a planned duration of at least 72 hours.

Exclusion Criteria:

* Magnetic resonance imaging planned, which would require removing the sensor less than 72 hours after installation;
* Patient whose death is expected within the next 72 hours.
* Patient included in the LOVIT study due to the theoretical risk of interference with blood glucose measurements with the CMS device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults hospitalized at the intensive care of the Centre hospitalier de l'Université de Montréal (CHUM), receiving an intravenous insulin infusion for more than 72 hours.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-07-27 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-01-11 (Estimated)

PRIMARY OUTCOMES:
To assess the validity of the Dexcom G6 CGM system measurements in IV insulin therapy patients hospitalized in the intensive care unit of the CHUM compared to the blood glucose measurements made using the Accuchek Inform II glucometer | 3-10 days

SECONDARY OUTCOMES:
To assess the validity of the Dexcom G6 CGM system measurements compared to the different methods of glucose measurement and different blood sources in intensive care | 3-10 days
  Comparing the Dexcom G6 CGM system measurements to the different methods of glucose measurement and different blood sources in intensive care:
  Portable glucometer, on capillary blood, Portable glucometer, on venous or arterial blood, Central laboratory analyzes on venous or arterial blood
Assess the validity of the Dexcom G6 CGM system measurements compared to the glucometer, according to the glucose concentrations measured: <4.0 mmol / L 4.0 - 10.0 mmol / L > 10.0 mmol / L | 3-10 days
To assess the validity of the Dexcom G6 CGM system measurements compared to the glucometer, according to the rate of change of glucose. | 3-10 days
Measure the influence of the patient's clinical characteristics (age, sex, weight, presence of diabetes, septic state and need for organ supports), and biochemical (hematocrit, acidosis, renal function) on the validity of CGM values. | 3-10 days
Assess the obstacles to the integration of the use of the CGM in the intensive care unit, namely the technical problems encountered and remote data management. | 3-10 days

CONTACTS AND LOCATIONS:
Overall Officials: Rémi Rabasa-Lhoret, MD, PhD, Principal Investigator — Institut de recherches cliniques de Montréal
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Canada